CLINICAL TRIAL: NCT06540534
Title: Comparison of Anesthetic and Analgesic Efficacy of Dexamethasone as an Adjuvant in Selective Trunk Block
Brief Title: Evaluation of Adjuvant Use in Selective Trunk Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: GaziosmanpasaTREHNA
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: Analgesia; Nerve Blocks; Postoperative Pain, Acute
Keywords: postoperative pain; postoperative analgesia; selective trunks block
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Dexamethasone; Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant-free selective trunks block (Active Comparator): In the selective trunk approach,Once the C6 and C5 ventral rami are identified at the level of the C7 transverse process, the probe will be slightly directed caudally to visualize the C6 ventral ramus. Caudal to the superior trunk, the middle trunk and the C8 ventral ramus will be visualized. The T1 ventral ramus can be seen on the 1st rib with the probe directed caudally. After administering 8 ml of the local anesthetic mixture to the lateral aspect of the superior trunk, the needle will be slightly withdrawn and directed towards the middle trunk where another 8 ml of the local anesthetic mixture will be administered. The probe will then be directed caudally to obtain an optimal view of the inferior trunk, and 9 ml of local anesthetic will be administered near the inferior trunk.
  In the control group, a total of 25 ml of local anesthetic mixture will be applied, consisting of 23 ml of 0.5% bupivacaine and 2 ml of 0.9% saline.
  Interventions: Procedure: kontrol group
- Adjuvant with selective trunks block (Active Comparator): In the selective trunk approach, Once the C6 and C5 ventral rami are identified at the level of the C7 transverse process, the probe will be slightly directed caudally to visualize the C6 ventral ramus. The probe will be used to scan until the area where the upper trunks of C5 and C6 are formed is observed. Caudal to the superior trunk, the middle trunk and the C8 ventral ramus will be visualized. After administering 8 ml of the local anesthetic mixture to the lateral aspect of the superior trunk, the needle will be slightly withdrawn and directed towards the middle trunk where another 8 ml of the local anesthetic mixture will be administered. The probe will then be directed caudally to obtain an optimal view of the inferior trunk, and 9 ml of local anesthetic will be administered near the inferior trunk.
  In the dexamethasone group, a total of 25 ml of local anesthetic mixture will be applied, consisting of 23 ml of 0.5% bupivacaine and 8 mg (2 ml of deksamethasone)
  Interventions: Procedure: Dexamethasone

INTERVENTIONS:
Procedure: Dexamethasone — In the adjuvan group (dexamethasone)group, a total of 25 ml of local anesthetic mixture will be applied, consisting of 23 ml of 0.5% bupivacaine and 2 ml of dexamethasone(8mg).
  Other Names: adjuvant
  Arms: Adjuvant with selective trunks block
Procedure: kontrol group — In the control group, a total of 25 ml of local anesthetic mixture will be applied, consisting of 23 ml of 0.5% bupivacaine and 2 ml of 0.9% saline.
  Other Names: salin group
  Arms: Adjuvant-free selective trunks block

SUMMARY:
"Evaluation of the Anesthetic and Analgesic Efficacy of Dexamethasone in Selective Trunk Blocks

DETAILED DESCRIPTION:
the investigators hypothesize that the perineural application of dexamethasone as an adjuvant in selective trunk block for upper extremity surgeries will accelerate the onset time of anesthesia and analgesia, provide significant anesthetic and analgesic effects, and prolong the duration of anesthesia and analgesia.

In recent years, the brachial plexus block, performed with various approaches, has been preferred over general anesthesia for upper extremity orthopedic surgeries due to its numerous advantages. It maintains the patient's consciousness and spontaneous respiration, reduces airway interventions, provides effective postoperative pain control, minimizes opioid-related side effects, limits surgery-related metabolic and endocrine changes, enables early discharge, and reduces treatment costs.

Selective trunk block offers rapid block onset and high success rates. The use of ultrasound in peripheral blocks has also reduced the risk of various complications (e.g., vascular injury). The selective trunk approach, as described by Manoj Kumar Karmakar in 2020, involves blocking the upper, middle, and lower trunks at the C7 transverse process level, resulting in sensory/motor block in all ipsilateral upper extremity dermatomes except T2. This study aims to compare the anesthetic and analgesic efficacy of dexamethasone as an adjuvant to bupivacaine in the selective trunk block approach.

Dexamethasone is a widely used glucocorticoid with anti-inflammatory, anti-toxic, and other effects. It has strong lipophilic properties, is soluble in fat, increases pH, facilitates the penetration of local anesthetics into nerve sheaths, and extends the duration of local anesthetic effects, as supported by various studies. Additionally, dexamethasone is commonly used in pain management for its neuromodulatory effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing upper extremity surgery with ASA (American Society of Anesthesiologists) classification I-II
* aged 18-65 years, and with a body mass index (BMI) between 18-35 kg/m² were included in the study.

Exclusion criteria:

* included ASA III-IV patients
* those who refuse the block
* pregnant and breastfeeding women
* individuals with severe lung disease
* contralateral diaphragm paralysis
* nerve injury secondary to trauma
* neuromuscular diseases,
* peripheral neuropathy
* bleeding diathesis
* history of anticoagulant use
* allergies to local anesthetics or dexamethasone
* uncontrolled diabetes mellitus
* morbid obesity with BMI >35 kg/m²
* severe cardiovascular, renal, or liver disease, and infections at the site where the nerve block is to be applied.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
onset times of motor and sensory blocks | first 30 minutes after the block aplication
  primary aim is to compare the effects of adding dexamethasone as an adjuvant to bupivacaine in selective trunk blocks on the onset times of motor and sensory blocks required for anesthesia.

SECONDARY OUTCOMES:
postoperative total motor block duration and analgesia duration. | within 24 hours after the surgery
  To compare the effects of dexamethasone as an adjuvant on postoperative total motor block duration and analgesia duration
first postoperative rescue analgesia | within 24 hours after the surgery hours
  To evaluate the time to the first postoperative rescue analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa Research and Education Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karmakar MK, Areeruk P, Mok LYH, Sivakumar RK. Ultrasound-Guided Selective Trunk Block to Produce Surgical Anesthesia of the Whole Upper Extremity: A Case Report. A A Pract. 2020 Jul;14(9):e01274. doi: 10.1213/XAA.0000000000001274. PMID 32909721
- [Result] Sivakumar RK, Samy W, Pakpirom J, Songthamwat B, Karmakar MK. Ultrasound-guided selective trunk block: Evaluation of ipsilateral sensorimotor block dynamics, hemidiaphragmatic function and efficacy for upper extremity surgery. A single-centre cohort study. Eur J Anaesthesiol. 2022 Oct 1;39(10):801-809. doi: 10.1097/EJA.0000000000001736. Epub 2022 Aug 11. PMID 35950709